CLINICAL TRIAL: NCT00602368
Title: Measurement of Digital Colposcopy for Fluorescence Spectroscopy of Cervical Intraepithelial Neoplasia: A Pilot Study
Brief Title: Digital Colposcopy in Finding Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000581286; BCCR-H03-61235 (Other: UBC-BCCA REB); P01CA082710 (NIH)
Record Dates: First submitted 2008-01-25; First posted 2008-01-28 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Histological Techniques; Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: histological technique
Other: laboratory biomarker analysis
Procedure: colposcopic biopsy
Procedure: colposcopy
Procedure: light-scattering spectroscopy
Procedure: loop electrosurgical excision procedure

SUMMARY:
RATIONALE: Diagnostic procedures, such as digital colposcopy, may help doctors find and diagnose cervical intraepithelial neoplasia.

PURPOSE: This clinical trial is studying digital colposcopy to see how well it works in finding cervical intraepithelial neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify potential improvements for a noninvasive method of diagnosing cervical dysplasia and neoplasia using digital colposcopy and fluorescence spectroscopic imaging.
* To measure fluorescence and reflectance images of the human cervix in vivo using digital colposcopy.
* To evaluate the effect of acetic acid on the image contrast obtained.
* To compare the device performance with colposcopic impression and histopathologic interpretation of tissue removed by standard loop electrosurgical excision procedure (LEEP).

OUTLINE: This is a multicenter study.

Participants undergo routine colposcopy as part of their regular colposcopic evaluation. The digital colposcope is used to take fluorescence and reflectance images of the vagina and cervix. Participants also undergo loop electrosurgical excision procedure (LEEP). The digital colposcopic images are compared with tissue removed during LEEP. Additional surrogate biomarkers under development are also measured using tissue samples removed during LEEP, such as quantitative histopathology measurements, DNA tests for the copy number changes, and tests for the incorporation of viral HPV DNA.

ELIGIBILITY:
Criteria:

Inclusion criteria:

* Included subjects will be ≥18 years old.
* Included subjects will not be pregnant.
* Included subjects will have a negative urine pregnancy test.
* Included subjects will be scheduled for colposcopy and/or LEEP treatment at the VGH Women's Clinic.
* Included subjects will indicate understanding of the study.
* Included subjects will provide informed consent to participate.

Exclusion criteria:

* Individuals <18 years old will be excluded.
* Pregnant individuals will be excluded.
* Individuals that have had an operation to remove their cervix will be excluded.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of digital colposcopy & fluorescence spectroscopy as a tool for early diagnosis of CIN | For length of study
  Measure normal and abnormal sites during colposcopy and compare this to pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Dianne M. Miller, M.D., Principal Investigator — British Columbia Cancer Agency, Vancouver General Hospital
Locations (1):
- BC Cancer Research Centre, Vancouver, British Columbia, Canada